CLINICAL TRIAL: NCT01549561
Title: Preventing Behavior and Health Problems in Foster Teens
Acronym: KEEP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KEEP2020172; R01DA020172 (NIH)
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Parent Management Training
Keywords: behavior problems; foster care; parent training; youth skills training
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Services As Usual (No Intervention): Foster care services as usual
- Parent and Youth Training (Experimental): 16 Weeks of Parent Training in group context with 5 to 10 relative and non-relative foster caregivers; Youth training with skills coaches
  Interventions: Behavioral: Parent Training; Behavioral: Youth Skills Training
- Parent Training (Experimental): 16 weeks of parent training with 5 to 10 relative and non-relative foster caregivers
  Interventions: Behavioral: Parent Training

INTERVENTIONS:
Behavioral: Parent Training — 16 weeks of parent training led by a trained group facilitator
  Other Names: Parent Management Training; KEEP
  Arms: Parent Training; Parent and Youth Training
Behavioral: Youth Skills Training — 16 weeks of one-on-one sessions with a trained youth skills coach
  Other Names: Skills Coaching
  Arms: Parent and Youth Training

SUMMARY:
The primary goal of this study is to test the efficacy of two levels of the KEEP intervention with adolescents and their foster and kin parents in the San Diego Child Welfare System.

DETAILED DESCRIPTION:
The cost of child welfare services in the U.S. has been estimated at $20 billion per year. During the past decade, the number of teenagers in foster care has nearly doubled. Numerous studies have documented that these adolescents are at high-risk for developing serious problems, including substance use, participation in health-risking sexual behaviors, involvement in the juvenile justice system, serious educational problems and school drop-out, failed placements/foster care "drift" and homelessness. Yet, there is little research on the characteristics of interventions that can be used to guide the improvement of services for this vulnerable population of youngsters. The proposed study extends our previous research with adolescents referred for serious behavioral and emotional problems and research with elementary-aged children in foster care to a test of the efficacy of a preventive intervention for adolescents placed with foster and kin care providers in the San Diego County Child Welfare System. Two hundred and forty adolescents and their foster/kin care providers will participate (i.e., 60 in a foster/kin parent training only condition, 60 in a parent training plus youth skill training condition, and 120 in a casework "as usual" control condition). In addition to testing the efficacy of the two levels of intervention, the investigators propose to examine the effects of the intervention on a set of youth behavioral and health-related outcomes. Parenting mediators to be tested include positive parenting, parental supervision, and non-harsh discipline. Youth mediators are social competence, commitment to school, and knowledge about norms related to health-risking behaviors including substance use and high-risk sexual behavior. In addition, theoretical hypotheses about the effects of early risk/adversity factors to youth outcomes will be examined, and an economic analysis will be conducted to examine the relative benefits and costs associated with the two levels of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any child between ages 12 and 16 years in relative or non-relative foster care

Exclusion Criteria:

* Only medically fragile children

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2006-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Reduction in child behavior problems as assessed by the Parent Daily Report (PDR) | Baseline, 6 Months, 12 Months, 18 Months

SECONDARY OUTCOMES:
Placement Disruptions from Foster Placement | 6 Months, 12 Months, 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Chamberlain, PhD, Principal Investigator — Oregon Social Learning Center
Locations (2):
- United States (2):
  - Child and Adolescent Services Research Center, San Diego, California
  - Oregon Social Learning Center, Eugene, Oregon

REFERENCES:
- [Background] Price, J., Chamberlain, P., Landsverk, J., & Reid, J. B. (2010). KEEP foster parent training intervention: Model description and effectiveness. Child and Family Social Work, 14, 233-242.